CLINICAL TRIAL: NCT05459870
Title: CAR-T Cells Targeting B Cell Related Autoimmune Diseases
Brief Title: CAR-T Cells Targeting Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Guilin Hospital of Chinese Traditional and Western Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-22010
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Autoimmune Diseases
Keywords: CAR-T; autoimmune disease; autoantibody; CD19; BCMA; CD138; BAFF-R
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4SCAR T Cell Therapy for autoimmune diseases (Experimental)
  Interventions: Biological: 4SCAR T cells

INTERVENTIONS:
Biological: 4SCAR T cells — Infusion of 4SCAR T cells at 10^6 cells/kg body weight via IV

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of CAR-T cell therapy in patients with autoimmune disease. Another goal of the study is to learn more about the safety and function of the CAR-T cells and their persistency in autoimmune disease patients.

DETAILED DESCRIPTION:
Autoimmune disease refers to the disease in which the immune system reacts to the host's own body and causes damage to tissues and organs. At present, the pathogenesis of various autoimmune diseases is still not well understood, but an imbalanced immune tolerance plays a key role in this process.

An ideal therapy to autoimmune disease should eradicate pathogenic autoimmune cells but retain the protective immunity. The chimeric antigen receptor-modified T (CAR-T) cell technology has proven to be highly effective in targeting B cell malignancies, and the treatment-induced B cell and antibody deficiencies have implications for treating autoantibody-related autoimmune diseases. Studies have shown that CAR-T cells targeting B cell surface molecules can kill autoreactive B lymphocytes in pemphigus vulgaris (PV) and systemic lupus erythematosus (SLE) patients. Thus, CAR-T cell technology targeting B cells has potential in treating autoimmune diseases including PV, SLE, autoimmune hemolytic anemia, Sjogren's syndrome etc..

CD19-specific CAR is based on activation of intracellular signalijng domains of T cells by the extracellular single chain variable fragment (scFv) antibody against CD19. The activated CAR-T cells can target and kill B cells. The investigation plans to use genetically modified T cells to express a 4th generation lentiviral anti-CD19 CAR with an inducible caspase 9 self-withdrawal gene (4SCAR) to increase the safety of this specific approach. Besides targeting CD19, specific CARs targeting other B cell surface molecules including BCMA, CD138, and BAFF-R will also be included in the treatment regimen. Based on accumulated experiences, the 4SCAR T cells have shown high safety profile without serious cytokine release syndrome (CRS) or neural toxicities in patients. Through this trial, the safety and long term efficacy of the B cell-specific 4SCAR T cell therapy will be evaluated, providing clinical evidence supporting the application of 4SCAR-T cell technology in the treatment of autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

1. age older than 18 years.
2. expression of B cell surface molecules.
3. the KPS score over 80 points, and survival time is more than 3 months.
4. greater than Hgb 80 g/L.
5. no contraindications to blood cell collection.

Exclusion Criteria:

1. accompanied with other active diseases and difficult to assess treatment response.
2. bacterial, fungal, or viral infection, unable to control.
3. living with HIV.
4. active HBV or HCV infection.
5. pregnant and nursing mothers.
6. under systemic steroid treatment within a week of the treatment.
7. prior failed CAR-T treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-31 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of 4SCAR T cells in patients with autoimmune diseases | 12 weeks
  Safety of 4SCAR T cells in patients with autoimmune diseases using CTCAE 5 standard to evaluate the level of adverse events

SECONDARY OUTCOMES:
B cell and immunoglobulin suppression activity of 4SCAR T cells in patients with autoimmune diseases | 1 year
  scale of CAR copies (for efficacy)
B cell and immunoglobulin suppression activity of 4SCAR T cells in patients with autoimmune diseases | 1 year
  immunoglobulin levels (for efficacy)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Guilin Hospital of Chinese Traditional and Western Medicine, Guilin, Guangxi

IPD SHARING:
Plan to Share IPD: No